CLINICAL TRIAL: NCT03800329
Title: Use of Remote Monitoring to Improve Physician Monitoring, Patient Satisfaction, and Predict Readmissions Following Cardiac Surgery
Brief Title: Remote Monitoring to Improve Physician Monitoring, Patient Satisfaction, and Predict Readmissions Following Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Snap40 Ltd. (Unknown)
Responsible Party: Principal Investigator, Jordan D. Miller, Ph.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-008249
Record Dates: First submitted 2018-08-14; First posted 2019-01-11 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Remote Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Snap40 Monitor (Active Comparator): Patients randomly assigned to wear the Snap40 monitor will wear the device for 48 hours following discharge from the hospital.
  Interventions: Device: Snap40 Monitor
- No Monitor (Placebo Comparator): Patients randomly assigned to not wear the Snap40 monitor will continue with their follow-up surgical care in the ordinary fashion.
  Interventions: Other: No Monitor

INTERVENTIONS:
Device: Snap40 Monitor — Non-invasive, wearable armband device used to measure change in systolic blood pressure, respiratory rate, heart rate, body temperature, movement, and oxyhemoglobin saturation and streams this information to a cloud-based storage system. Patients will complete a questionnaire.
  Arms: Snap40 Monitor
Other: No Monitor — Patients will be discharged in the ordinary manner, without the Snap40 monitor. Patients will complete a questionnaire.
  Arms: No Monitor

SUMMARY:
This study is designed to determine the perceived value of continuous remote monitoring to surgeons and surgical patients at Mayo Clinic in Rochester, MN, and determine whether algorithms can be generated to predict risk of readmission following discharge. This initial study will be conducted through the Department of Cardiovascular Surgery.

DETAILED DESCRIPTION:
The overall aim of this project is to determine the perceived utility and benefit to use of remote monitoring technology in patients being discharged following cardiac surgery at Mayo Clinic in Rochester, MN. The investigators also aim to determine whether machine learning algorithms can predict readmission following cardiac surgery in these patients, which the investigators believe will benefit patients in future studies.

ELIGIBILITY:
Target accrual: 100 patients

Subject population (children, adults, groups): adults undergoing coronary bypass surgery at Mayo Clinic in Rochester, MN

Inclusion Criteria:

* Patients undergoing isolated coronary artery bypass graft (CABG) surgery
* Must be undergoing the procedure at Mayo Clinic in Rochester, MN
* Must be greater than or equal to 40 years of age

Exclusion Criteria:

* Under 40 years of age
* Concomitant additional surgical procedure (e.g., CABG + valve replacement)
* Patients with implantable pacemakers/defibrillators
* Patients that find the device too uncomfortable to wear for 48 hours

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Physician satisfaction in the use of remote monitoring technology. | 48 hours
  Physician satisfaction survey measure the utility and benefit to the use of remote monitoring technology in patients being discharged following cardiac surgery at Mayo Clinic in Rochester, MN.

SECONDARY OUTCOMES:
Patient satisfaction in the use of remote monitoring technology. | 48 hours
  Patient satisfaction survey measures the utility and benefit to the use of remote monitoring technology in patients being discharged following cardiac surgery at Mayo Clinic in Rochester, MN.

OTHER OUTCOMES:
Algorithms useful in prediction of readmission following cardiac surgery | 48 hours
  Measure data collected via machine learning algorithms to predict readmission following cardiac surgery in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan D Miller, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials